CLINICAL TRIAL: NCT00095628
Title: A Phase 2 Study of SB-715992 in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: SB-715992 in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03091; PHL-031; 6803; N01CM62203 (NIH)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — ispinesib; CK0238273

ARMS (1):
- Treatment (ispinesib) (Experimental): Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ispinesib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: ispinesib — Given IV
  Other Names: CK0238273; SB-715992
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well SB-715992 works in treating patients with recurrent or metastatic head and neck cancer. Drugs used in chemotherapy, such as SB-715992, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the antitumor activity of SB-715992 in recurrent and/or metastatic squamous cell carcinoma of the head and neck using objective response rates (partial and complete responses).

SECONDARY OBJECTIVES:

I. To determine the duration of objective response, rate and duration of stable disease, progression-free, median and overall survival rates of SB-715992 in recurrent and/or metastatic squamous cell carcinoma of the head and neck.

II. To document the safety and tolerability of SB-715992 in recurrent and/or metastatic squamous cell carcinoma of the head and neck.

III. To characterize the population pharmacokinetic (PK) parameters of SB-715992 including an assessment of significant covariates on SB-715992 PK and an assessment of the potential relationships between the pharmacokinetics of SB-715992 and relevant safety and efficacy endpoints.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell carcinoma of the head and neck that is recurrent or metastatic; with the exception of the nasopharynx, all primary sites (including oral cavity, oropharynx, hypopharynx, and larynx) will be eligible; MedDRA disease terms:

  * Oral neoplasms NOS, 10031008
  * Oropharyngeal cancer recurrent, 10031098
  * Hypopharyngeal cancer recurrent, 10021044
  * Laryngeal cancer recurrent, 10023828
  * Maxillofacial sinus neoplasm, 10026956
  * Head and neck, 90002024
* Patients may have had a maximum of one prior chemotherapy regimen for recurrent or metastatic disease; patients may enter this study and receive SB-715992 as their first-line therapy for recurrent and/or metastatic disease; prior platinum-based chemotherapy delivered concurrently with radiotherapy, or prior platinum-based induction chemotherapy, is allowed; there must be at least a 4 week interval between any chemotherapy (6 weeks for nitrosoureas or mitomycin C), radiotherapy or surgery and study enrollment; exceptions may be made however, for low dose, non-myelosuppressive radiotherapy - please contact the Principal Investigator (Dr. E. Winquist) PRIOR to registration if questions arise about the interpretation of this criterion; for patients who received local therapy prior to study entry, there must be either progression of measurable disease documented within the treatment field, or must have measurable disease outside the treatment field prior to study entry
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Life expectancy of greater than 12 weeks.
* ECOG performance status 0,1, or 2
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 3.0 X institutional upper limit of normal (=< 5.0 X if liver metastases)
* Creatinine =< 1.5 X institutional upper limit of normal
* Peripheral neuropathy may be no greater than grade 1
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of SB-715992 will be determined following review of their use by the TREATING RESPONSIBLE investigator; patients receiving nonprohibited medications or substances known to interact with CYP450 isoenzymes may be eligible but should be monitored carefully; questions about eligibility related to concommitant use of medications should be discussed with the Principal Investigator
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring INR. If medically appropriate and treatment available, the investigator may also consider switching these patients to LMW heparin, where an interaction with SB-715992 is not expected
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with non-squamous cell carcinomas of the head and neck or nasopharyngeal cancer
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from AEs due to agents administered more than 4 weeks earlier
* Patients may not have received any other investigational agents within 28 days of study entry
* Patients may not receive other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study
* The following lists of medications/substances are moderate to significant inhibitors/inducers of CYP3A4 that, if administered concomitantly with SB-715992, may alter study drug exposure; the use of these medications/substances within 14 days (>= 6 months for amiodarone) prior to the administration of the first dose of SB-715992 through discontinuation from the study is prohibited

  * Inhibitors of CYP3A4:

    * Antibiotics: clarithromycin, erythromycin, troleandomycin
    * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200 mg/day), voriconazole
    * Antidepressants: nefazodone, fluovoxamine
    * Calcium channel blockers: verapamil, diltiazem
    * Miscellaneous: amiodarone*, grapefruit juice, bitter orange

      * Use of amiodarone within 6 months prior to the administration of the first dose of SB-715992 is prohibited
  * Inducers of CYP3A4:

    * Anticonvulsants: phenytoin, carbamazepine, Phenobarbital, oxcarbazepine
    * Antibiotics: rifampin, rifabutin, rifapentine
    * Miscellaneous: St. John's wort, modafinil
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SB-715992
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because SB-715992 is a mitotic inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SB-715992, breastfeeding should be discontinued if the mother is treated with SB-715992

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winquist, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ispinesib)
Started | 21
Completed | 20
Not Completed | 1
Not completed — Disease progression prior to treatment | 1

BASELINE CHARACTERISTICS:
Population: A total of 21 patients were enrolled onto the study. One patient was ineligible due to disease progression prior to treatment. So a total of 20 evaluable patients were analyzed
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: participants] | 60 [41 to 75]
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Region of Enrollment [Number; unit: participants]
  Canada | 18
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity of SB-715992 Using Objective Response Rates (Partial and Complete Responses)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesion
Time Frame: Up to 18 months
Population: 20 eligible patients were analyzed
Measure: Number; unit: participants
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Duration of Objective Response
Description: as for outcome 1
Time Frame: Up to 18 months
Population: Data were not collected because 0 participants showed a response.
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Clinical and Objective Stable Disease
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease.
Time Frame: Up to 18 months
Measure: Number; unit: participants
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 20
participants | 5

4. Secondary Outcome: Median Overall Survival of SB-715992
Description: Overall survival is defined as the time from enrolment until death due to any cause. The Kaplan-Meier method was used to estimate overall survival.
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 20
months | 3.5 [2.8 to 7.8]

5. Secondary Outcome: Median Time to Progression
Description: Time to progression (TTP) is defined as the time from enrolment onto the study until progression or death. The Kaplan-Meier method was used to estimate TTP.
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 20
months | 1.4 [1.3 to 2.3]

6. Other Pre Specified Outcome: 1 Year Overall Survival
Description: as for outcome 4
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ispinesib)
Number analyzed (Participants) | 20
percentage of participants | 20 [8.3 to 48.1]

ADVERSE EVENTS:
Arm/Group | Treatment (Ispinesib)
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ispinesib) (N=20)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Leukopenia (Investigations) | 1 (1) — White blood count decreased
Neutropenia (Investigations) | 1 (1) — Neutrophil count decreased
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Edema face (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Injury to superior vena cava (Injury, poisoning and procedural complications) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ispinesib) (N=20)
Neutropenia (Investigations) | 14 — Neutrophil count decreased
Leukopenia (Investigations) | 15 — White blood count decreased
Nausea (Gastrointestinal disorders) | 9
Lymphopenia (Investigations) | 9 — Lymphocyte count decreased
Anemia (Blood and lymphatic system disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 6
Fatigue (General disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Injection site reaction (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less